CLINICAL TRIAL: NCT06570551
Title: Continuous Glucose Monitoring System Use in Pediatric Patients with Diabetes
Status: Completed | Type: Observational
Sponsor: Sinocare (Industry)
Responsible Party: Sponsor
Other Study IDs: NPI031-CIP-005
Record Dates: First submitted 2024-08-12; First posted 2024-08-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 2-5 year old participants: Wear the investigational device continuously for 15 days.
  Interventions: Device: i3 CGM(continuous glucose monitor)
- 6-17 year old participants: Wear the investigational device continuously for 15 days.
  Interventions: Device: i3 CGM(continuous glucose monitor)

INTERVENTIONS:
Device: i3 CGM(continuous glucose monitor) — The i3 CGM consists of a Sensor Pack (including probe, iCGM-S3), a Transmitter Pack (iCGM-t3), and an application (iCGM-APP (released version: V02)).application (i3 CGM App). The user can view their glucose data on the i3 CGM App running on a compatible mobile device.

SUMMARY:
To verify and evaluate the efficacy and safety of i3 CGM system manufactured by Changsha Sinocare Inc. for continuous or regular monitoring of interstitial fluid glucose level in pediatric patients with diabetes.

DETAILED DESCRIPTION:
This clinical investigation is of a multi-center and self-controlled design.

This clinical investigation is planned to be conducted in 3 study sites, with a total of 78 subjects to be enrolled, of which no fewer than 15 cases are aged 2-5 years old, and no fewer than 60 cases are aged 6-17 years old. This clinical investigation is to verify the safety and efficacy of the investigational device. Referring to the number of pediatric patients with diabetes in the 3 study sites, it is expected that about 20 subjects will be enrolled in each site every month, and it will take about 2 months to close the site. This clinical investigation is expected to be completed in about 6 months from the first participant recruited.

The real-time glucose values measured by CGM system on the left and right abdomen are compared with the venous blood glucose value (EKF value) measured by EKF analyzer, respectively, and the consistency rate is analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 (inclusive) - 18 years (exclusive);
* Clinically diagnosed with diabetes;
* Being willing to wear the device continuously for 15 days and conduct blood collection for blood glucose testing in accordance with the requirements of this protocol;
* Body weight not less than 10.0 kg;
* Consent to participate in this clinical investigation, and sign the Informed Consent Form (ICF).

Exclusion Criteria:

* Need to undergo magnetic resonance imaging (MRI) during the clinical investigation;
* Diffuse subcutaneous nodules;
* Acute complications of diabetes;
* Abnormal coagulation function (coagulation cannot be too quick or too slow); the criteria for judging abnormalities are: The activated partial thromboplastin time (APTT) is higher than 1.5 times the upper limit of normal value or lower than the lower limit of normal value; or The prothrombin time (PT) is higher than 1.5 times the upper limit of normal value or lower than the lower limit of normal value
* Participation in other clinical investigations within the past 1 month;
* Where the investigator does not consider the patient suitable for enrollment.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 2-17 year old patients with diabetes mellitus.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2024-03-30 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
Accuracy | 0-15 days
  percentage of i3 CGM values in the measuring range less than 4.4 mmol/L(80 mg/dL) within ± 1.1 mmol/L(20 mg/dL) of the EKF control.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Hunan Children's Hospital, Changsha, Hunan
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - Women and Children's Hospital of Ningbo University, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No